CLINICAL TRIAL: NCT00233740
Title: The Cordis Protection From Pulmonary Embolism With the Permanent OptEase™ Filter - A Post Marketing Surveillance Study (PROOF Study)
Brief Title: Protection From Pulmonary Embolism With the Permanent OptEase™ Filter (PROOF)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P02-7001
Record Dates: First submitted 2005-10-04; First posted 2005-10-06 (Estimated); Last update posted 2008-08-05 (Estimated); Status verified 2008-08

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: OPTEASE Vena Cava Filter

SUMMARY:
The main objective of this study is to monitor the safety and effectiveness of the OptEase™ Permanent Vena Cava (IVC) Filter

ELIGIBILITY:
Inclusion Criteria:

* · Pulmonary thromboembolism when anticoagulants are contraindicated.

  * Failure of anticoagulant therapy in thromboembolic diseases.
  * Emergency treatment following massive pulmonary embolism where anticipated benefits of conventional therapy are reduced.
  * Chronic, recurrent pulmonary embolism where anticoagulant therapy has failed or is contraindicated.

Exclusion Criteria:

* · Patients with risk of septic embolism.

  * Patients with uncontrolled infectious disease.
  * Patients with an IVC diameter > 30 mm.
  * Patients contraindicated for procedures under fluoroscopy.
  * Patients with demonstrated hypersensitivity to one or more of the components of the OptEase™ filter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2003-09; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
The co-primary endpoints are migration of the OptEase™ IVC filter as determined by abdominal x-ray at 1-month post-implantation and symptomatic thrombosis at 1-month post-implantation. Migration is defined as > 2 cm movement in either cranial or caudal

SECONDARY OUTCOMES:
To assess major adverse event rates related to the filter or filter procedure, up to 6-month follow-up, in aggregate and individually. Major adverse events are defined as 1) death, 2) pulmonary embolism, 3) symptomatic thrombosis, 4) caval penetration
To assess the longer-term stability of the filter defined by the lack of migration as seen on abdominal x-ray at 6-month post-implantation. Migration is defined as > 2 cm movement in either cranial or caudal direction as seen on abdominal x-ray compar
To assess the clinical success of the filter up to 6-month follow-up. Clinical success is defined as the absence of symptomatic pulmonary embolism (PE) evaluated clinically at post-implantation, 1- and 6-months post-implantation.
To assess the technical success of the filter up to 6-month follow-up. Technical success is defined as the filter successfully deployed at the intended site in the IVC with the correct orientation.
To assess significant tilting (> 15° off the axis of the IVC) up to 6-month follow-up.
To assess filter fracture up to 6-month follow-up.
Procedure-related bleeding (defined as requiring transfusion or > 3 gm decrease in hemoglobin).

CONTACTS AND LOCATIONS:
Overall Officials: Peter Weidenfeld, MD, Principal Investigator — Sunrise Hospital and Medical Center

REFERENCES:
- [Result] Ziegler JW, Dietrich GJ, Cohen SA, Sterling K, Duncan J, Samotowka M. PROOF trial: protection from pulmonary embolism with the OptEase filter. J Vasc Interv Radiol. 2008 Aug;19(8):1165-70. doi: 10.1016/j.jvir.2008.04.020. Epub 2008 Jun 27. PMID 18656008